CLINICAL TRIAL: NCT06416371
Title: Retinal Vessel Leakage in Cerebral Small Vessel Disease: a Sub-study of the Mild Stroke Study 3
Brief Title: Retinal Vessel Leakage in Cerebral Small Vessel Disease
Status: Recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: AC24000
Record Dates: First submitted 2024-01-15; First posted 2024-05-16 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Small Vessel Diseases; Lacunar Stroke; Vascular Dementia
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Stroke, Lacunar; Dementia, Vascular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Fundus fluorescein angiography, with ultrawide field retinal imaging — Intravenous injection of sodium fluorescein for angiography of retinal blood vessels

SUMMARY:
The goal of this observational study is to learn about leakage from retinal vessels in cerebral small vessel disease. The main questions it aims to answer are:

* Does retinal vessel leakage occur in cerebral small vessel disease?
* If it does, is the severity of retinal vessel leakage similar to the severity of cerebral small vessel disease generally?

Participants will be tested using fluorescein angiography. This involves an intravenous injection of fluorescent dye, and is a very sensitive way to find leakage from retinal blood vessels.

Participants will have already had brain scans and other examinations and tests to measure the severity of their cerebral small vessel disease. Our new retinal images will complement the information from these previous tests.

DETAILED DESCRIPTION:
Cerebral small vessel disease (SVD) is a common cause of stroke and dementia. The molecular causes are unclear, limiting new therapies. Breakdown of the blood-brain barrier (BBB) is characteristic and may damage brain tissue. However, specialist MRI scans to measure BBB breakdown are expensive and time-consuming.

In contrast, measuring leakage from retinal blood vessels is relatively simple. The blood-retina barrier is very similar to the BBB, and SVD is likely to damage retinal and brain blood vessels in the same way. If so, then retinal angiography could be used to study SVD pathogenesis and measure the effect of new treatments with much greater resolution and lower cost than MRI.

We have three aims:

1. Test the feasibility of fluorescein angiography in people with SVD
2. Discover if retinal vessel leakage occurs people with SVD
3. Discover whether the severity of retinal vessel leakage is associated with clinical features of SVD

We will recruit participants from a well-established cohort of people with SVD - the Mild Stroke Study 3 (MSS3).

ELIGIBILITY:
Inclusion Criteria:

* Membership in the Mild Stroke Study 3 cohort
* Contrast enhanced MRI within 12 months
* Clear optical media in both eyes, as assessed by study investigator
* Best corrected visual acuity (near vision) ≥N36

Exclusion Criteria:

* Any condition known to cause retinal leakage (i.e., worse than background diabetic retinopathy, retinal vein occlusion, active uveitis, wet age-related macular degeneration, malignant hypertension)
* Previous treatment for retinal leakage (retinal laser, intravitreal anti-VEGF)
* Recent eye surgery
* Shallow anterior chambers as assessed by torch test
* Pregnancy, renal failure
* Severe dementia
* Known allergy to fluorescein
* History of allergy such as food or drug induced urticaria or history of bronchial asthma
* Any other severe or acute medical or psychiatric conditions
* Inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults >18 years old with mild ischaemic stroke with a modified Rankin scale (mRS) greater or equal to 2 at recruitment presenting to Edinburgh/Lothian stroke services.
  For details see Clancy, et al (2021) Rationale and design of a longitudinal study of cerebral small vessel diseases, clinical and imaging outcomes in patients presenting with mild ischaemic stroke: Mild Stroke Study 3. European Stroke Journal 6:81-88. https://doi.org/10.1177/2396987320929617
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Retinal vessel leakage by automated segmentation | within one angiogram
  The presence and severity of retinal vessel leakage will be measured for each eye in terms of change in pixel brightness over the duration of the angiogram.
Retinal vessel leakage by manual grading | within one angiogram
  The presence and severity of retinal vessel leakage will be measured using an manual ordinal grading scale

SECONDARY OUTCOMES:
Baseline blood-brain barrier breakdown | Within one MRI scan
  BBB breakdown is measured by MRI in terms of image enhancement after intravenous gadolinium
White matter hyperintensity (WMH) volume adjusted for brain volume | Within one MRI scan
  This is measured from the most recent structural MRI scan
Change in white matter hyperintensity (WMH) volume adjusted for brain volume | Difference in MRI scans up to 5 years prior
  This is measured by comparing the most recent structural MRI scan with the baseline structural MRI scan
Fazekas score | Within one MRI scan
  This is measured from the most recent structural MRI scan
Change in Fazekas score | Difference in MRI scans up to 5 years prior
  This is measured by comparing the most recent structural MRI scan with the baseline structural MRI scan
Baseline average leakage in white matter hyperintensities | Within one MRI scan
  BBB breakdown is measured by MRI in terms of image enhancement after intravenous gadolinium
Baseline average leakage in deep grey matter | Within one MRI scan
  BBB breakdown is measured by MRI in terms of image enhancement after intravenous gadolinium
Baseline number of leakage hotspots | Within one MRI scan
  BBB breakdown is measured by MRI in terms of image enhancement after intravenous gadolinium

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clancy U, Garcia DJ, Stringer MS, Thrippleton MJ, Valdes-Hernandez MC, Wiseman S, Hamilton OK, Chappell FM, Brown R, Blair GW, Hewins W, Sleight E, Ballerini L, Bastin ME, Maniega SM, MacGillivray T, Hetherington K, Hamid C, Arteaga C, Morgan AG, Manning C, Backhouse E, Hamilton I, Job D, Marshall I, Doubal FN, Wardlaw JM. Rationale and design of a longitudinal study of cerebral small vessel diseases, clinical and imaging outcomes in patients presenting with mild ischaemic stroke: Mild Stroke Study 3. Eur Stroke J. 2021 Mar;6(1):81-88. doi: 10.1177/2396987320929617. Epub 2020 Jun 5. PMID 33817338
- [Background] MacCormick IJ, Maude RJ, Beare NA, Borooah S, Glover S, Parry D, Leach S, Molyneux ME, Dhillon B, Lewallen S, Harding SP. Grading fluorescein angiograms in malarial retinopathy. Malar J. 2015 Sep 24;14:367. doi: 10.1186/s12936-015-0897-7. PMID 26403288